CLINICAL TRIAL: NCT06837558
Title: Predictors of Bone Mineral Density in Lupus Nephritis Activity
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ammar ahmed ammar, Assiut university, Assiut University
Other Study IDs: Bone mass in lupus nephritis
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Bone Mineral Density and Lupus Nephritis Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- lupus nephritis in active form: 1. Full history taking suggestion of SLE according to WHO criteria
  2. Complete physical examination (as blood pressure, pulse, chest, heart, abdomen examinations, lower limbs edema, puffiness of eyes)
  3. Investigations: including the different following modalititis
  A. Laboratory investigations include:
  1. Complete blood picture, PT PC INR, RBS Kidney function tests, eGFR Urine analysis, 24 hours' protein in urine
  2. Specific laboratory investigations for SLE and lupus nephritis: ANA,AntiDsDNA,C3,C4 Laboratory investigations of Bone mineral density predictors Ca, phosphorus, PTH, vitamin D (OH), Alkaline phosphatase, Fibroblast Growth Factor 23 (FGF 23)
  B. Imaging studies:
  1 - Abdominal ultrasound 2- chest x-ray 3- Echocardiography (in lupus nephritis with acti
  Interventions: Diagnostic Test: fibroblast growth factor 23
- lupus nephritis in inactive form: 1- Full history taking suggestion of SLE according to WHO criteria 2- Complete physical examination (as blood pressure, pulse, chest, heart, abdomen examinations, lower limbs edema, puffiness of eyes) 3- Investigations: including the different following modalititis A. Laboratory investigations include: 1- Complete blood picture, PT PC INR, RBS Kidney function tests, eGFR Urine analysis, 24 hours' protein in urine 2- Specific laboratory investigations for SLE and lupus nephritis: ANA,AntiDsDNA,C3,C4 Laboratory investigations of Bone mineral density predictors Ca, phosphorus, PTH, vitamin D (OH), Alkaline phosphatase, Fibroblast Growth Factor 23 (FGF 23) B. Imaging studies: 1 - Abdominal ultrasound 2- chest x-ray 3- Echocardiography (in lupus nephritis with acti
  Interventions: Diagnostic Test: fibroblast growth factor 23

INTERVENTIONS:
Diagnostic Test: fibroblast growth factor 23 — Investigations: including the different following modalititis
  A. Laboratory investigations include:
  1. Complete blood picture, PT PC INR, RBS Kidney function tests, eGFR Urine analysis, 24 hours' protein in urine
  2. Specific laboratory investigations for SLE and lupus nephritis: ANA,AntiDsDNA,C3,C4
  3. Laboratory investigations of Bone mineral density predictors Ca, phosphorus, PTH, vitamin D (OH), Alkaline phosphatase, Fibroblast Growth Factor 23 (FGF 23)
  B. Imaging studies:
  1 - Abdominal ultrasound 2- chest x-ray 3- Echocardiography (in lupus nephritis with activity form) 4- DEXA bone scan
  C. Invasive modality:
  Renal biopsy of Patients with SLE with lupus nephritis
  Other Names: DEXA bone scan

SUMMARY:
Our aim in this study is Correlation of histopathology of renal biopsy in SLE with lupus nephritis patients versus predictors of bone mineral density in active and inactive lupus nephritis

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an autoimmune disorder characterized by multisystem damage, leading to significant health issues [1]. There is growing concern over the adverse effects of medications used to treat SLE and the potential long-term complications [2]. Lupus nephritis (LN) is a severe and frequently manifestation of SLE, associated with significant morbidity and mortality [3-5]. Research indicates that female patients with SLE are at a higher risk of developing reduced bone mineral density (BMD) [6-9]. Moreover, women exhibit a high prevalence of osteoporosis and osteoporotic fractures [10]. Osteoporosis is a common and serious complication of SLE, contributing to increased morbidity and mortality rates [11, 12]. there is a notable gap in the literature regarding osteoporosis prevalence among LN patients. Risk factors such as glucocorticoid therapy, early menopause, and low calcium and vitamin D intake are known to contribute to bone loss [13-16], yet the specific risk factors associated with osteoporosis in LN patients vary by country, indicating a need for further research in this area. The pathophysiology of bone mineral density (BMD) reduction in Systemic Lupus Erythematosus (SLE), particularly in relation to lupus nephritis (LN) activity, is multifactorial and complex. The mechanisms behind this association involve immune system dysregulation, chronic inflammation, steroid use, kidney dysfunction, and alterations in mineral metabolism (17)

ELIGIBILITY:
Inclusion Criteria:

The patients with lupus nephritis based on KDIGO over 18 years and less than 60 years The patient diagnosed as SLE with lupus nephritis and in active form. The patient diagnosed as SLE with lupus nephritis and without active criteria The patient consent.

Exclusion Criteria:

Patients with SLE and also diagnosed as end stage renal disease on regular hemodialysis

* Association of another autoimmune as rheumatoid arthritis
* Association of HCV, HBV
* Association of diabetes mellitus or malignancy
* Patient had history of vitamin D supplementation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients attending outpatient clinics and inpatient of Internal Medicine department of Assiut University Hospital .The study will be done on total of 100 patients with SLE divided into:
  (A): 50 Patients with SLE with lupus nephritis with activity (B): 50 Patients with SLE with lupus nephritis without activity
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of histopathology of renal biopsy in SLE with lupus nephritis patients versus predictors of bone mineral density in active and inactive lupus nephritis | From 1/4/2025 to 1/4/2027
  All patients in this study will be subjected to:
  1. Full history taking suggestion of SLE according to WHO criteria
  2. Complete physical examination (as blood pressure, pulse, chest, heart, abdomen examinations, lower limbs edema, puffiness of eyes)
  3. Investigations: including the different following modalititis
  A. Laboratory investigations include:
  1. Complete blood picture, PT PC INR, RBS Kidney function tests, eGFR Urine analysis, 24 hours' protein in urine
  2. Specific laboratory investigations for SLE and lupus nephritis: ANA,AntiDsDNA,C3,C4
  3. Laboratory investigations of Bone mineral density predictors Ca, phosphorus, PTH, vitamin D (OH), Alkaline phosphatase, Fibroblast Growth Factor 23 (FGF 23)
  B. Imaging studies:
  1 - Abdominal ultrasound 2- chest x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Nashwa Moustafa Abdel Monem Azoz, assistant professor nephrology, Study Chair — Assiut university hospital internal medicine

REFERENCES:
- [Background] Siegel CH, Sammaritano LR. Systemic Lupus Erythematosus: A Review. JAMA. 2024 May 7;331(17):1480-1491. doi: 10.1001/jama.2024.2315. PMID 38587826